CLINICAL TRIAL: NCT00832481
Title: Comparison of the Effects of Repaglinide and Metformin on Glucose Excursions in Newly Diagnosed Type 2 Diabetes Patients in China
Brief Title: Comparison of the Effects of Repaglinide and Metformin on Glucose Excursions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Chinese PLA General Hospital, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: NovoNorm 301 Chunlin Li
Record Dates: First submitted 2009-01-29; First posted 2009-01-30 (Estimated); Last update posted 2009-08-25 (Estimated); Status verified 2009-08

CONDITIONS: Type 2 Diabetes
Keywords: Repaglinide; Metformin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — repaglinide; Tablets; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Repaglinide,tablet (Active Comparator)
  Interventions: Drug: Repaglinide
- Metformin, tablet (Active Comparator)
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Repaglinide — Repaglinide (NovoNorm®): 0.5 mg/tablet, 1.0 mg/tablet
  Other Names: Repaglinide (NovoNorm®): 0.5 mg/tablet
  Arms: Repaglinide,tablet
Drug: Metformin — 2 mg/tablet Metformin (Glucophage®): 0.5 g/tablet
  Other Names: Metformin (Glucophage®): 0.5 g/tablet
  Arms: Metformin, tablet

SUMMARY:
This is a 17 week, randomized, single center, open-label, parallel-group study to compare glucose excursions and other efficacy and safety parameters of repaglinide thrice daily or metformin thrice daily in newly diagnosed type 2 diabetes subjects in China.

DETAILED DESCRIPTION:
This is a 17 week, randomized, single center, open-label, parallel-group study to compare glucose excursions and other efficacy and safety parameters of repaglinide thrice daily or metformin thrice daily in newly diagnosed type 2 diabetes subjects in China.

Eligibility for participation will be determined by medical history, physical examination, and laboratory results obtained during a screening visit (see trail population). About 60 patients with newly diagnosed (within 6 months) type 2 diabetes and both insulin and oral antidiabetic drugs (OAD) naïve will be include in this study. All subjects will be given informed consent before starting any examination and test. Then the 24h blood glucose of each patient will be recorded by utilizing continue glucose monitor system (CGMS). Besides that, the following data of all subject will be collected: HbA1c, Fasting blood glucose, 2h postprandial blood glucose, fasting lipid profile, 2h postprandial lipid profile, fasting uric acid, 2h postprandial uric acid, fasting insulin and proinsulin, 2h postprandial insulin and proinsulin, fasting C peptide, 2h postprandial C peptide, fasting glucagon, 2h postprandial glucagon.

After baseline data are collected, eligible subjects will be randomized into each group at a 2:1 ratio (40 for repaglinide and 20 for metformin). IVGTT and hyperinsulinemic-euglycemic clamp will be done to 20 patients in repaglinide group and 10 patients in metformin group (less than 20% drop-off rate is acceptable for this study). Follow that, all patients will start to receive either repaglinide thrice daily (immediately before breakfast lunch, and dinner) or metformin thrice daily (after breakfast, lunch and dinner). The initial repaglinide doses will be based on HbA1c levels on the day of randomization (0.5 mg tid for HbA1c < 8% and 1 mg tid for HbA1c ≥ 8%); the initial dosage for metformin will be 0.5 g tid and this dosage will be kept until the end of this study.

Treatment diaries will be asked for every subject to record glucose levels (7 times per day and 2 days per week for the first three weeks, then 7 times per day and 1 day per week until the end of this study), diet and exercise, stress situation, hypoglycemic symptoms and so on. All patients will be followed by visiting clinic every week for the first three weeks, but only patients in repaglinide group will be titrated their doses. Dose adjustment should be aimed at achieving the following glycemic targets: fasting blood glucose: 4.4 - 6.0 mmol/L, 2h post prandial glucose 4.4 - 8.0 mmol/L. If above glycaemic target has not been achieved, repaglinide dose should be adjusted for every week (see Schematic diagram of trial design). The adjustment of repaglinide doses is based on the mean of blood glucose recorded in subject diaries. The doses of repaglinide before each meal may be different, depending on the recorded blood glucose concentrations. After three weeks titration for repaglinide (maximal dosage for repaglinide is 2 mg tid), the patients in this group will keep the optimal dosage for the next 12 weeks. Clinic visit will be conducted every four weeks after the period of dosages titration to collect information, such as hypoglycemia, adverse events and fasting blood glucose.

Complicated examinations will be repeated again after above 12 weeks treatments for both groups, including physical examination, electrocardiogram (ECG), CGMS, fasting and 2h post prandial glucose, concentration of insulin, proinsulin, C peptide, glucagon, uric acid and so on. IVGTT and hyperinsulinemic-euglycemic clamp will be repeated only for subjects who did that at the beginning of study. Data will be collected and analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent obtained before any trial-related activities. (Trial- related activities are any procedure that would not have been performed during normal management of the subject.)
2. Ages between 20-90 years
3. BMI between 18.5 and 30 kg/m2
4. Newly diagnosed type 2 diabetes. Type 2 diabetes is in accordance with WHO criteria 1999
5. The history of diabetes less than 6 months
6. HbA1c <10%.
7. Only on diet and/or exercise, OAD or insulin naïve subjects

Exclusion Criteria:

1. Any history of OAD or insulin therapy preceding this trial.
2. Type 1 diabetic subjects, including LADA
3. Pregnant, breast-feeding or the intention of becoming pregnant or not using adequate contraceptive measures (adequate contraceptive measures are sterilisation, IUD, oral contraceptives or barrier methods) before and/or during the trial.
4. Impaired hepatic function (ALT > 2.5 times upper limit of local laboratories normal ranges)
5. Impaired renal function, defined as serum creatinine ≥ 1.5 mg/dl.
6. Use of systemic or inhaled glucocorticoids or other medication known to interfere with glucose metabolism.
7. Recently had acute diabetic complications
8. Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation.
9. Recently had operation, injury, inflammation and other stress conditions.
10. Recently had cardiac disease as following:

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-10 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
To investigate the effects of monotherapy of either repaglinide or metformin on glucose excursion after 3 months treatment in newly diagnosed type 2 diabetes patients in China | from Jan.01 2009 to Oct.30,2009

CONTACTS AND LOCATIONS:
Overall Officials: Chunlin Li, M.D&Ph.D, Principal Investigator — PLA General Hospital
Locations (1):
- PLA General Hospital, Beijing, Beijing Municipality, China